CLINICAL TRIAL: NCT00449449
Title: A Randomised, Open, Controlled, Parallel Group, Multi-Centre Phase II Clinical Study of Lidocain Pertubation as Treatment for Couples With Unexplained Infertility
Brief Title: A Phase II Clinical Study of Lidocain Pertubation as Treatment for Couples With Unexplained Infertility
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Isifer AB (Industry)
Collaborators: Karolinska Institutet (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISI-03-1
Record Dates: First submitted 2007-03-17; First posted 2007-03-20 (Estimated); Last update posted 2007-03-20 (Estimated); Status verified 2007-03

CONDITIONS: Infertility
Keywords: Pertubation, tubal flushing, intrauterine insemination.
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Pertubation with Lidocain Solution

SUMMARY:
The study tested the hypothesis that a pertubation with a lidocain solution will enhance pregnancy rate.

DETAILED DESCRIPTION:
In a prospective study, patients were randomized during a clomiphene citrate stimulated cycle to either pertubation with low-dose lidocain or no pertubation before insemination.

ELIGIBILITY:
Inclusion Criteria:

* Female,
* 20-40 years of age,
* If presence of peritoneal endometriosis they must be of minimal or mild without adhesions (verified by laparoscopy),
* Normal menstruation cycle,
* Male partner 20-70 years of age,
* Male partner,
* Normal sperm sample within 5 years (>20x106/mL, total sperm count >30x106, normal morphology 5%),
* Duration of infertility more than one year,
* Signed informed consent

Exclusion Criteria:

* Treatment with NSAID, corticosteroids or other drugs, which can cause an increased risk of infection,
* Clinical signs of PID,
* Known hypersensitivity to local anesthetics,
* Non-patent fallopian tubes,
* Pathological uterine cavity,
* Pathological PCT, myoma > 2 cm diameter,
* Any disease or laboratory finding considered of importance by the investigator not to include the patient

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 330
Dates: Start 2003-09; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
clinical pregnancy

SECONDARY OUTCOMES:
Pregnancy rate measured by Serum-HCG day 17 after IUI

CONTACTS AND LOCATIONS:
Overall Officials: Greta Edelstam, Md. PhD, Principal Investigator — Department of Obstetrics and Gynecology, Karolinska University Hospital at Huddinge, S-141 86 Stockholm, Sweden
Locations (1):
- 1. Department of Obstetrics and Gynecology, Karolinska University Hospital at Huddinge, Stockholm, Stockholm County, Sweden

REFERENCES:
- [Derived] Edelstam G, Sjosten A, Bjuresten K, Ek I, Wanggren K, Spira J. A new rapid and effective method for treatment of unexplained infertility. Hum Reprod. 2008 Apr;23(4):852-6. doi: 10.1093/humrep/den003. Epub 2008 Feb 15. PMID 18281242